CLINICAL TRIAL: NCT02535897
Title: The Effects of an Insulinotropic Protein-carbohydrate Beverage on L- Carnitine Absorption and Muscle Carnitine Uptake
Brief Title: Protein Ingestion and Muscle Carnitine Uptake
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: G26062012 BMS
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Muscle, Skeletal
MeSH Terms: interventions — Carbohydrates; Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CON (Placebo Comparator): 500 ml of flavoured water
  Interventions: Dietary Supplement: Flavoured water
- CHO (Active Comparator): 500 ml of flavoured water containing 80 g carbohydrate
  Interventions: Dietary Supplement: Flavoured water + carbohydrate
- CHO-PRO (Active Comparator): 500 ml of flavoured water containing 40 g carbohydrate and 40 g whey protein
  Interventions: Dietary Supplement: Flavoured water + carbohydrate + protein

INTERVENTIONS:
Dietary Supplement: Flavoured water
  Arms: CON
Dietary Supplement: Flavoured water + carbohydrate
  Arms: CHO
Dietary Supplement: Flavoured water + carbohydrate + protein
  Arms: CHO-PRO

SUMMARY:
The purpose of this study is to assess the effects of a protein-carbohydrate beverage on the absorption of an orally ingested bolus of L-carnitine, compared to flavoured water and carbohydrate-only controls, and to determine whether increasing plasma carnitine availability can impact upon insulin-stimulated muscle carnitine uptake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Body mass index of 18-25 kg/cm2

Exclusion Criteria:

* Unhealthy
* Smoker
* Taking any medication that interferes with skeletal muscle metabolism

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Muscle carnitine uptake | 180 minutes
  Change in forearm carnitine uptake (measured using arterialised-venous - venous balance technique) in response to intervention.